CLINICAL TRIAL: NCT01357070
Title: Does Broccoli Sprout Consumption Result in Plasma Sulforaphane Levels That Can Attenuate Leukocyte Activation Ex-vivo in Healthy Human Volunteers?
Brief Title: Effect of Broccoli Sprout on Blood Levels of Sulforaphane to Reduce Responsiveness of Immune System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2-bao
Record Dates: First submitted 2011-05-17; First posted 2011-05-20 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Healthy Volunteers
Keywords: white blood cell; broccoli; P38 Map Kinase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brocco-sprout homogenate (Active Comparator)
  Interventions: Dietary Supplement: Brocco-sprout homogenate
- Alfalfa sprout homogenate (Sham Comparator)
  Interventions: Dietary Supplement: Alfalfa sprout homogenate

INTERVENTIONS:
Dietary Supplement: Brocco-sprout homogenate — Participants will be asked to orally consume on three consecutive days a brocco-sprout homogenate (70g dry weight).
  Arms: Brocco-sprout homogenate
Dietary Supplement: Alfalfa sprout homogenate — Participants will be asked to orally consume on three consecutive days an alfalfa sprout homogenate.
  Arms: Alfalfa sprout homogenate

SUMMARY:
The investigators suggest that inducing anti-oxidant enzymes indirectly may be an effective means of providing vascular protection.

Sulforaphane, a naturally occurring compound found in green vegetables (including broccoli, brussel sprouts and cauliflower) is able to protect against cell inflammatory stress by inducing a number of anti-oxidant molecules. Targeted studies on the consumption of broccoli and related vegetables have been shown to be associated with reduced risk of coronary artery disease.

In the present study the investigators want to test whether the consumption of a "broccoli smoothie" containing sulforaphane can protect white blood cells from becoming activated in the presence of an experimental stress and how long this protective effect lasts for. To do this, the investigators will be analysing inflammatory changes in blood samples taken at different times during the study.

DETAILED DESCRIPTION:
Atherosclerosis is the disease process that leads to hardening of the arteries which causes them to become narrowed. This occurs because fat is first deposited on the inside walls of the arteries, then becomes hardened by fibrous tissue and calcium deposition forming a semi-hardened accumulation of material known as plaque. As this plaque grows, it narrows the channel within the artery and causes a reduction in blood and oxygen supply to the affected organ - such as the heart and brain. The investigators now understand that this process is caused by inflammation and activation of the immune cells over a period of time. It has been proposed that targeting these immune cells and reducing the levels of immune activation can protect against cardiovascular diseases.

Previously it has been observed that consumption of fruit and vegetables rich in anti-oxidants can confer a protective effect against cardiovascular diseases. The use of anti-oxidants experimentally has shown protective benefits against activation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ years
* Able to commit for the two week duration of the trial

Exclusion Criteria:

* Age <18 years
* Pregnancy
* Vegetarian
* History of allergy
* Current smoker or smoking cessation within the last 3 months
* Current use of inhaled, topical or systemic corticosteroids or within the last 2 weeks
* Current use of non-steroidal anti-inflammatory use or within the last 1 week
* Current use of nutritional or multivitamin supplements
* Current participation in any other Randomised controlled trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Resistance of leucocytes to inflammatory activation following an experimental stress | 24 hours after consumption of the third homogenate
  Participants will consume a brocco-sprout homogenate. Blood will be sampled for intracellular markers of leukocyte stress after ex-vivo stimulus with Phorbol ester / Tumour Necrosis Factor alpha. The following parameters will be recorded.
  1. Reactive oxygen species detection using aminophenylfluoresceine dye
  2. p38 MAP kinase induction
  3. NF-kB induction

CONTACTS AND LOCATIONS:
Overall Officials: Paul C Evans, BSc MSc PhD, Principal Investigator — Imperial College London
Locations (1):
- Cardiovascular Medicine Research Unit, Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Clinical Study Report: DOI:10.4172/2472-1921.100060 — https://clinical-nutrition.imedpub.com/consumption-of-broccoli-sprouts-attenuatesintracellular-p38-map-kinase-and-reactiveoxygen-species-proinflammatory-activationin-hum.php?aid=21325 — RESULTS REPORT